CLINICAL TRIAL: NCT03102762
Title: Intracavernosal Injection of Botulinum Toxin Type A in the Treatment of Erectile Dysfunction (Phase 2 Study)
Brief Title: Botulinum Toxin for Erectile Dysfunction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hussein Ghanem, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1232017
Record Dates: First submitted 2017-03-28; First posted 2017-04-06 (Actual); Results first posted 2019-12-05 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Sexual Dysfunction; Erectile Dysfunction
Keywords: Erectile dysfunction; Botulinum toxin A; Botox
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Erectile Dysfunction | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective, randomized double blind placebo control ( RDBPC) study.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botulinum Toxin Type A (BTX-A) Group (Experimental): Experimental: BTX-A Group The treatment group, 35 patients, will be injected with 100 units BTX-A one day following penile colour Doppler assessment.
  Interventions: Drug: Botulinum Toxin Type A
- Placebo Group (Placebo Comparator): Saline Group:
  The control group, 35 patients, will be injected with 1 ml normal saline one day following penile colour Doppler assessment.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Drug: Botulinum Toxin Type A The treatment group will be injected with 100 units BTX-A one day following penile colour doppler assessment.
  Arms: Botulinum Toxin Type A (BTX-A) Group
Drug: Normal saline — The treatment group will be injected with 1 ml normal saline one day following penile colour doppler assessment.
  Arms: Placebo Group

SUMMARY:
To evaluate the safety and efficacy of intra-cavernosal Botulinum toxin injection as an alternative line of treatment in patients with erectile dysfunction - not responding to oral PDE5i - through cavernosal smooth muscle relaxation.

DETAILED DESCRIPTION:
The initial Phase 1 study demonstrated safety and efficacy of Botulinum toxin type A in the treatment of Erectile dysfunction in a small randomized controlled trial of 24 men.

The investigators conduct a phase 2 trial to confirm the initial results in a larger group of men.70 males will be included in the study. The participants will be subjected for full history taking, general and genital examination. Penile duplex will be performed to assess a vascular etiology before the treatment and 2 weeks later. The patients will be randomized into a treatment group (35 patients) and a control group (35 patients).

All patients will sign an informed consent. The treatment group will be injected IC with a trimix solution (20 ug alprostadil + 1 mg phentolamine + 30 mg papaverine) for color Doppler assessment, followed, next day by 50 units of BTX-A. The control group will be injected with the trimix solution during penile color Doppler assessment followed next day with a normal saline injection. The erection hardness score (EHS) will be assessed during the Doppler exam.

Procedure: At least 1 day after the penile color Doppler test, the patient is placed in the supine position flaccid and stretched penile length and girth would be measured from tip of the penis to the pubic bone will be done. A rubber band will be applied to the base of the penis. The skin will be prepped with alcohol swabs followed by the IC injection of 100 units of BTX-A. Direct pressure will be applied for 2 minutes. The rubber band will be removed after 15 minutes.

Patients and controls will fill the Sexual Health Inventory for men (SHIM) questionnaire and answer the the Sexual Encounter Profile questions 1 and 2 (SEP 2 & SEP 3), and the global assessment question (GAQ) before and 4 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 70 males will be included in the study recruited from Andrology, Sexology & STD's outpatient clinic, Kasr El Aini Hospitals, Cairo University, complaining of ED.
* Unable to develop erections sufficient for intercourse.
* Failing to respond to first line and second line treatments for Erectile Dysfunction with surgery as the only remaining treatment option.
* Age between 18 to 80 years.

Exclusion Criteria:

- Significant cardiovascular disease interfering with sexual activity

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Islam M Fathy, MD, Study Director — Cairo University; Abdelrahman A Hassan, Msc, Study Director — Cairo University
Locations (1):
- Department of Andrology, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghanem H, Soliman I, AbdulHamid M, et. PS-08-016 Can intracavernosal botulinum toxin injection salvage vascular erectile dysfunction patients not responding to oral and intracavernous therapy? A pilot study. May 2016. Volume 13, Issue 5, Supplement 2, Page S116.
- See also: Botulinum Toxin Type A and Erectile Dysfunction (Phase 1 study) — https://clinicaltrials.gov/ct2/show/record/NCT02584686

RESULTS

PARTICIPANT FLOW:
Groups:
- BTX-A Group: Experimental: BTX-A Group The treatment group, 35 patients, will be injected with 100 units BTX-A one day following penile colour Doppler assessment.
  Botulinum Toxin Type A: Drug: Botulinum Toxin Type A The treatment group will be injected with 100 units BTX-A one day following penile colour doppler assessment.
- Placebo Group: Saline Group:
  The control group, 35 patients, will be injected with 1 ml normal saline one day following penile colour Doppler assessment.
  Normal saline: The treatment group will be injected with 1 ml normal saline one day following penile colour doppler assessment.
Period: Overall Study
Arm/Group | BTX-A Group | Placebo Group
Started | 35 | 35
Completed | 34 | 35
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: One patient was dropped out from the treatment group 6 weeks after of BTX injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | BTX-A Group | Placebo Group | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.26 (7.8) | 56 (9.12) | 55.13 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 35 | 35 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Egyptian | 35 | 35 | 70
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Right (PSV R) and Left (PSV L) Cavernosal Artery Mean PSV Before Treatment
Description: Baseline mean Peak systolic velocity (PSV) in the Cavernosal arteries, on color Doppler examination, in the patient and control groups.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | BTX-A Group | Placebo Group
Number analyzed (Participants) | 35 | 35
cm/sec
  PSV R | 34.52 (12.15) | 30.85 (15.26)
  PSV L | 34.33 (11.21) | 31.73 (15.97)

2. Primary Outcome: Right (PSV R) and Left (PSV L) Cavernosal Artery Mean PSV After Treatment
Description: Cavernosal artery mean peak systolic velocity (PSV) after treatment, on color Doppler examination, in the patient and control groups.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | BTX-A Group | Placebo Group
Number analyzed (Participants) | 35 | 35
cm/sec
  PSV R | 45.68 (13.27) | 31.67 (15.67)
  PSV L | 46.015 (13.03) | 32.09 (16.47)

3. Secondary Outcome: SHIM Score Before Treatment
Description: Assessment of the Sexual Health Inventory for men (SHIM) questionnaire before treatment for both groups. It is a questionnaire that helps asses if the patient has erectile dysfunction (ED) and assesses its degree. Results range from 1 to 25. A score of 1-7 denotes Severe ED, 8-11 Moderate ED, 12-16, Mild to Moderate ED, 17-21 Mild ED, 22-25 No ED.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BTX-A Group | Placebo Group
Number analyzed (Participants) | 35 | 35
score on a scale | 5.4 (1.67) | 5.69 (1.08)

4. Secondary Outcome: SHIM Score After Treatment
Description: Assessment of the Sexual Health Inventory for men (SHIM) questionnaire after treatment for both groups. It is a questionnaire that helps to asses if the patient has erectile dysfunction (ED) and to assess its degree. Results range from 1 to 25. A score of 1-7 denotes Severe ED, 8-11 Moderate ED, 12-16, Mild to Moderate ED, 17-21 Mild ED, 22-25 No ED.
  Minimum value is 1, Maximum value is 25, the higher the score the better is the outcome.
Time Frame: 2 weeks after injection.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BTX-A Group | Placebo Group
Number analyzed (Participants) | 35 | 35
score on a scale | 6.66 (2.17) | 6.11 (2.82)

5. Secondary Outcome: SHIM Score After Treatment
Description: Assessment of the Sexual Health Inventory for men (SHIM) questionnaire after 6 and 12 weeks of both groups. It is a questionnaire that helps to asses if the patient has erectile dysfunction (ED) and to assess its degree. Results range from 1 to 25. A score of 1-7 denotes Severe ED, 8-11 Moderate ED, 12-16, Mild to Moderate ED, 17-21 Mild ED, 22-25 No ED.
  Minimum value is 1, Maximum value is 25, the higher the score the better is the outcome.
Time Frame: 6 and 12 weeks after injection.
Population: One patient was dropped out after 2 weeks of injection from the BTX-A Group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Botulinum Toxin Type A (BTX-A) Group | Placebo Group
Number analyzed (Participants) | 34 | 35
score on a scale
  6 weeks after injection | 9.97 (5.92) | 5.77 (1.82)
  12 weeks after injection | 8.26 (4.07) | 5.57 (1.399)

6. Secondary Outcome: Penile Size Before Treatment
Description: Measurement of penile length before treatment:
  Flaccid, stretched and erect penile length.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | BTX-A Group | Placebo Group
Number analyzed (Participants) | 35 | 35
cm
  Flaccid penile length | 10.17 (1.73) | 10.99 (2.49)
  Stretched penile length | 13.36 (1.8) | 13.4 (2.58)
  Erect penile length | 14.17 (1.72) | 14.01 (2.56)

7. Secondary Outcome: Penile Size After Treatment
Description: Measurement of penile length after treatment.
Time Frame: 2 weeks after injection.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | BTX-A Group | Placebo Group
Number analyzed (Participants) | 35 | 35
cm
  After 2 weeks flaccid | 10.46 (1.8) | 11.01 (2.52)
  After 2 weeks stretched | 13.41 (1.78) | 13.4 (2.58)
  After 2 weeks erect | 14.26 (1.66) | 14.03 (2.57)

8. Secondary Outcome: Penile Size After Treatment
Description: Measurement of penile length after treatment.
Time Frame: 6 and 12 weeks after injection.
Population: One patient was dropped out from the treatment group after 2 weeks injection.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Botulinum Toxin Type A (BTX-A) Group | Placebo Group
Number analyzed (Participants) | 34 | 35
cm
  After 6 weeks flaccid | 10.54 (1.83) | 10.99 (2.49)
  After 6 weeks stretched | 13.46 (1.81) | 13.4 (2.58)
  After 12 weeks flaccid | 10.46 (1.74) | 10.99 (2.49)
  After 12 weeks stretched | 13.44 (1.79) | 13.4 (2.58)

9. Secondary Outcome: Intra-vaginal Latency Time Before Treatment
Description: Measurement of the duration of intercourse from intromission to ejaculation before treatment.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | BTX-A Group | Placebo Group
Number analyzed (Participants) | 35 | 35
Participants
  IVLT less than 1 minutes | 12 | 9
  IVLT from 1 to 3 minutes | 13 | 18
  IVLT more than 3 minutes | 10 | 8

10. Secondary Outcome: Intra-vaginal Latency Time After Treatment
Description: Measurement of the duration of intercourse from intromission to ejaculation after treatment.
Time Frame: 2 weeks after injection.
Measure: Count of Participants; unit: Participants
Arm/Group | BTX-A Group | Placebo Group
Number analyzed (Participants) | 35 | 35
Participants
  After 2 weeks IVLT less than 1 minute | 12 | 8
  After 2 weeks IVLT between 1 to 3 minutes | 13 | 18
  After 2 weeks IVLT more than 3 minutes | 10 | 9

11. Secondary Outcome: Intra-vaginal Latency Time After Treatment
Description: Measurement of the duration of intercourse from intromission to ejaculation after treatment.
Time Frame: 6 and 12 weeks after injection.
Population: One patient was dropped out from the treatment group after 2 weeks injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Botulinum Toxin Type A (BTX-A) Group | Placebo Group
Number analyzed (Participants) | 34 | 35
Participants
  After 6 weeks IVLT less than 1 minute | 9 | 8
  After 6 weeks IVLT between 1 to 3 minutes | 15 | 19
  After 6 weeks IVLT more than 3 minutes | 10 | 8
  After 12 weeks IVLT less than 1 minute | 9 | 8
  After 12 weeks IVLT between 1 to 3 minutes | 14 | 19
  After 12 weeks IVLT more than 3 minutes | 11 | 8

ADVERSE EVENTS:
Time Frame: Adverse effects were collected at 2, 6 and12 weeks for each patient throughout the study.
Groups:
- BTX-A Group: Experimental: BTX-A Group The treatment group, 80 patients, will be injected with 100 units BTX-A one day following penile colour Doppler assessment.
  Botulinum Toxin Type A: Drug: Botulinum Toxin Type A The treatment group will be injected with 100 units BTX-A one day following penile colour doppler assessment.
- Placebo Group: Saline Group:
  The control group, 80 patients, will be injected with 1 ml normal saline one day following penile colour Doppler assessment.
  Normal saline: The treatment group will be injected with 1 ml normal saline one day following penile colour doppler assessment.
Arm/Group | BTX-A Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT03102762/Prot_SAP_000.pdf